CLINICAL TRIAL: NCT04038268
Title: Criteria Used by Health Professionals on the Selection of Allergen Immunotherapy in Real Clinical Practice: an International E-survey
Brief Title: Criteria Used by Health Professionals on the Selection of Allergen Immunotherapy in Real Clinical Practice
Acronym: CHOICE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0361
Record Dates: First submitted 2019-07-12; First posted 2019-07-30 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Allergen Immunotherapy
Keywords: Immunotherapy; Real Clinical Practice; Respiratory disease; Aeroallergens; IgE-dependent hypersensitivity
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Adults and children, males and females, with IgE mediated pollen, house dust mites, animal dander and moulds respiratory allergy who will initiate aeroallergen AIT, either SCIT, SLIT-drops or SLIT-tablets according to real life clinical standards of practice
- Prescribers: Doctors who are currently prescribing AIT as part of their regular clinical practice

SUMMARY:
Background : Allergen Immunotherapy (AIT) is the only etiological treatment for allergic respiratory diseases. In order to improve the competence on the use of AIT, it is important to extend the investigator's knowledge on its use in routine clinical practice, outside the experimental setting of clinical trials, in real life population of patients receiving AIT.

Objective: To evaluate the clinical criteria used by treating clinicians and by the patients themselves, when establishing AIT as treatment in a patient with respiratory disease caused by an IgE-dependent-hypersensitivity to aeroallergens Methods: In 6 country (Denmark, France, Germany, Norway, Spain & Sweden), the national coordinator will be directly responsible for selection of Survey Doctor's participants (Investigators).

During 12 months:

* Firstly, each investigator will complete the Survey Doctor, online, on SurveyMonkey platform to explain what are the key drivers in Allergen Immunotherapy (AIT) selection (Doctors' Questionnaire, DQ).
* On the other hand, at each AIT prescription to a patient, doctors will complete the Survey Patient, on the same platform, to explain how and why they have chosen this type of AIT (Patients' Questionnaire, PQ).

ELIGIBILITY:
Inclusion criteria:

* Patients with IgE mediated respiratory allergy
* Patients who will initiate any type of aeroallergen AIT according to real life clinical standards of practice
* Any type of aeroallergen for AIT will be included : pollen, house dust mite, animal, dander, moulds
* Patient who is under the care of the Doctor participating in the survey

Exclusion criteria:

* Patients who refuse to give their informed consent
* Food immunotherapy
* Venom Immunotherapy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with IgE mediated hypersensitivity to aeroallergens who will initiate AIT, either SCIT, SLIT-drops or SLIT-tablets according to real life clinical standards of practice
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical criteria in AIT | 1 day
  Clinical criteria used by treating clinicians and by the patients themselves, when establishing AIT as treatment in a patient with respiratory disease. These are called "drivers of prescription".
  caused by an IgE-dependent-hypersensitivity to aeroallergens Among the different criteria selected by participants, order of priority of AIT drivers will be established

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Demoly, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC